CLINICAL TRIAL: NCT06529835
Title: A Comparison of NeuroSpan Bridge, NeuraGen Nerve Guide, and Nerve Autograft for Peripheral Nerve Repair (NeuroSpan-1)
Brief Title: A Comparison of NeuroSpan Bridge, NeuraGen Nerve Guide, and Nerve Autograft for Peripheral Nerve Repair
Acronym: NeuroSpan-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auxilium Biotechnologies (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUX-NS-001
Record Dates: First submitted 2024-07-22; First posted 2024-07-31 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Peripheral Nerve Injuries
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Intervention Model Description: A total of 80 subjects will be enrolled and randomized using a 1:1 ratio.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding will occur to the subject and the blinded assessor. The blinded assessor will remain blinded from the device that was implanted. For subjects, blinding will be accomplished by informing subjects during the consent process that they may or may not also receive a secondary procedure in which they could have an incision in their leg that is not dependent on the device in which they are randomized to receive. Blinding will be assessed by the use of blinding assessment to both the assessor at the patient at the 12 month follow-up visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- NeuroGen Nerve Guide (Active Comparator): The control arm will comprise of subjects requiring injury repair of 0.5-1.0cm. These subjects will receive the NeuraGen Nerve Guide.
  Interventions: Device: NeuroSpan Bridge; Device: NeuroGen Nerve Guide
- Nerve Autograft (Active Comparator): The control arm will comprise of subjects requiring injury repair of 1.1-3.0cm. These subjects will receive the Nerve Autograft.
  Interventions: Device: NeuroSpan Bridge; Device: Nerve Autograft

INTERVENTIONS:
Device: NeuroSpan Bridge — The implant is used to connect peripheral nerve discontinuities. It is designed to be an interface between the nerve and surrounding tissue and to create a conduit for axonal growth across a nerve gap.
  The NeuroSpan Bridge is a novel scaffold to support regeneration that mimics the natural bio- architecture, providing multiple channels that are strictly linear so that axonal position is accurately maintained across the full length of the scaffold - over any length - to re-enter the distal nerve stump.
Device: NeuroGen Nerve Guide — The NeuraGen Nerve Guide is a resorbable implant for the repair of 0.5-1.0cm peripheral nerve discontinuities. NeuraGen Nerve Guide provides a protective environment for peripheral nerve repair after injury. It is designed to be an interface between the nerve and surrounding tissue and to create a conduit for axonal growth across a nerve gap. The semi-permeable type 1 collagen membrane allows for controlled resorption, appropriate nutrient diffusion and retention of representative Nerve Growth Factor.
  Arms: NeuroGen Nerve Guide
Device: Nerve Autograft — A nerve autograft is a surgical procedure that involves transplanting a segment of a patient's own sensory nerve tissue to repair a damaged peripheral nerve injury measuring 1.1-3.0cm. It is designed to be an interface between the nerve and surrounding tissue and to create a conduit for axonal growth across a nerve gap
  Arms: Nerve Autograft

SUMMARY:
This is a multicenter, prospective, randomized, subject and evaluator blinded clinical trial to asses the efficacy of Auxilium's NeuroSpan Bridge.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 with upper or lower extremity nerve injury with a gap of 0.5 to 3.0 cm.
2. Nerve diameter at injury site ≤3mm.
3. Nerve injury location is the arm from the shoulder to the wrist, including the hand or the leg from the hip to the ankle including the foot.
4. For Motor Nerve Injuries: Distance from site of injury to the nearest innervated muscle: ≤100mm
5. For Sensory and Mixed Nerve injuries: Distance from the site of injury to the nearest sensory nerve target: ≤250mm
6. Repair must take place within 3 months from injury
7. No contraindications to surgical repair (e.g., risk of concurrent infection, dog bite)

Exclusion Criteria:

1. Previous history of nerve repair attempt at the treated nerve.
2. Concurrent disease that reduces nerve regeneration: diabetes, previous diagnosis of non-traumatic peripheral neuropathy, chemotherapy treatment, other causes of peripheral neuropathy.
3. Allergy to Bovine products such as Bovine Collagen Nerve Cuff.
4. Pregnancy or planning to become pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy- Static two-point discrimination (s2PD) measured at 12 months. | 12 months
  This endpoint will examine the change in Static two-point discrimination (s2PD) measured at 12 months.
Safety- Complications and adverse events including infections, inflammation, tissue rejections, neuroma formation, chronic pain, and device malfunctions occurring between the treatment procedure and the 12-month follow-up visit. | 12 months
  This endpoint will examine complications and adverse events including infections, inflammation, tissue rejections, neuroma formation, chronic pain, and device malfunctions occurring between the treatment procedure and the 12-month follow-up visit.

SECONDARY OUTCOMES:
Motor function assessed by the British Medical Research Council grading system (categories 0, 1, 2, 3, 4, 5) at 12 months. | 12 months
  This endpoint will examine motor function assessed by the British Medical Research Council grading system (categories 0, 1, 2, 3, 4, 5) at 12 months.
Sensory function assessed by the British Medical Research Council grading system at 12 months. | 12 months
  This endpoint will examine sensory function assessed by the British Medical Research Council grading system at 12 months.
Moving 2 Point Discrimination test (m2PD) in the target digit at 12 months. | 12 months
  This endpoint will examine Moving 2 Point Discrimination test (m2PD) in the target digit at 12 months.
The summary score from the Disabilities of the Arm Shoulder and Hand (DASH) questionnaire at 12 months. | 12 months
  This endpoint will examine the summary score from the Disabilities of the Arm Shoulder and Hand (DASH) questionnaire at 12 months.
  The Disabilities of the Arm Shoulder and Hand (DASH) is a 30-item patient-reported outcome measure utilized to assess symptoms and function of the entire upper extremity. It is scored using the 5-point Likert-Scale measuring from "1" (lowest level of difficulty or severity) to 5" (highest level of difficulty or severity) based on the patient's reported ability to conduct the activities or tasks. A higher score indicates greater disability.
The summary score from the Disabilities of the Arm Shoulder and Hand (DASH) Work Module at 12 months. | 12 months
  This endpoint will examine the summary score from the Disabilities of the Arm Shoulder and Hand (DASH) Work Module at 12 months.
  The Disabilities of the Arm Shoulder and Hand (DASH) Work Module is a 4 question patient-reported outcome measure utilized to assess the impact of the patients arm, shoulder, or hand problem on the patients ability to work. It is scored using the 5-point Likert-Scale measuring from "1" (lowest level of difficulty or severity) to 5" (highest level of difficulty or severity) based on the patient's reported ability to conduct the activities or tasks. A higher score indicates greater disability.
The summary score from the Disabilities of the Arm Shoulder and Hand (DASH) Sports/Performing Arts Module at 12 months. | 12 months
  This endpoint will examine the summary score from the Disabilities of the Arm Shoulder and Hand (Dash) Sports/Performing Arts Module at 12 months.
  The Disabilities of the Arm Shoulder and Hand (DASH) Sports/Performing Arts Module is a 4 question patient-reported outcome measure utilized to assess the impact of the patients arm, shoulder, or hand problem on their ability to play a musical instrument, participate in sport or both. It is scored using the 5-point Likert-Scale measuring from "1" (lowest level of difficulty or severity) to 5" (highest level of difficulty or severity) based on the patient's reported ability to conduct the activities or tasks. A higher score indicates greater disability.

OTHER OUTCOMES:
Decrease in Surgery time between NeuroSpan Bridge vs. Nerve Autograft. | 12 months
  This clinical measure will examine the decrease in Surgery time between NeuroSpan Bridge vs. Nerve Autograft.
Comparison in Surgery time between NeuroSpan Bridge vs. NeuraGen Nerve Guide. | 12 months
  This clinical measure will examine the comparison in Surgery time between NeuroSpan Bridge vs. NeuraGen Nerve Guide.
Changes in Numerical Rating Scale (NRS) pain scores from baseline. | 12 months
  This clinical measure will examine changes in Numerical Rating Scale (NRS) pain scores from baseline. Numerical Rating Scale (NRS) is a pain scale that measures a patient's pain intensity or other features. Patients are asked to circle the number between 0 and 10 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the 10 represents 'the worst pain ever possible'.
Hospital/Outpatient center readmission rates within 30 days of surgery. | 30 days
  This clinical measure will examine the Hospital/Outpatient center readmission rates within 30 days of surgery

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCSF Orthopedic Institute, San Francisco, California
  - Medstar Union Memorial Hospital- The Curtis National Hand Center, Baltimore, Maryland
  - NYU Langone Orthopedic Center, New York, New York
  - OSU Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - The San Antonio Orthopaedic Group (TSAOG Orthopaedics), San Antonio, Texas